CLINICAL TRIAL: NCT02279004
Title: A Prospective Study of Plasma Genotyping as a Noninvasive Biomarker for Genotype-directed Cancer Care
Status: Recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Damon Runyon Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Julia K. Rotow, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 14-147
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: NSCLC; Melanoma
Keywords: Plasma Genotyping; NSCLC; Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell-free plasma DNA (cfDNA) derived from tumor cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Newly Diagnosed Patients: Newly diagnosed patients with advanced NSCLC or melanoma with complete or planned tissue genotyping.
- Acquired Resistance Patients: NSCLC patients with a known EGFR mutation or other targetable mutation and acquired resistance to initial kinase inhibitor therapy.
- Known Genotype Patients: NSCLC patients with a known genomic alteration detectable by ddPCR-based plasma genotyping and planned to start a new line of therapy.
- Advanced NSCLC: Advanced NSCLC patients with a biopsy planned for tissue genotyping.

SUMMARY:
Tumor genotyping has become an essential biomarker for the care of advanced lung cancer and melanoma, and is currently used to identify patients for treatment with targeted kinase inhibitors like erlotinib and vemurafenib. However, tumor genotyping can be slow and cumbersome, and is limited by availability of tumor biopsy tissue for testing. The aim of this study is to prospectively evaluate a blood-based genotyping tool that can quantify the presence of oncogenic mutations (EGFR, KRAS, BRAF) in patients with lung cancer and melanoma. This assay is being studied both as a diagnostic tool for classifying patient genotype, and a serial measurement tool for quantification of response and progression on therapy.

ELIGIBILITY:
Inclusion Criteria

To participate in this study a participant must meet the eligibility of one of the following cohorts:

Cohort 1: Cancers beginning initial treatment

* One of the following diagnoses:

  * Cohort 1A (CLOSED):

    ---Advanced non-squamous NSCLC (including adenosquamous)
  * Cohort 1B:

    * Stage II-III non-squamous NSCLC (including adenosquamous)
    * Stage IIIB-IV melanoma
* Patient must be planned to begin initial therapy, or completely resected before or after receiving adjuvant therapy
* For patients with NSCLC, EGFR and KRAS genotype may be known or unknown
* For patients with melanoma, BRAF and NRAS genotype may be known or unknown
* For patients without tumor genotyping, there must be a plan for genotyping including either:

  * Archived tumor tissue available and planned for genotyping
  * A biopsy at some future time is anticipated and will be available for genotyping

Cohort 2: Cancers with acquired resistance to targeted therapy

* One of the following diagnoses:

  * Cohort 2A (CLOSED):

    ---Advanced NSCLC harboring a known EGFR mutation
  * Cohort 2B:

    * Advanced NSCLC harboring a targetable genotype other than EGFR
    * Advanced melanoma harboring a known tumor genotype
* Clinical determination of progression targeted therapy, as evidence by plans to start a new systemic treatment regimen, or obtain a biopsy to plan a new treatment regimen

  * New systemic treatment regimen planned OR
  * Re-biopsy for resistance genotyping planned
* Note, date of targeted therapy start and clinical progression must be provided

Cohort 3: Cancers with a known genotype starting palliative systemic therapy

Cohort 3A (CLOSED):

* Advanced NSCLC harboring one of the following mutations:

  * EGFR exon 19 deletion
  * EGFR L858R
  * EGFR T790M
  * KRAS G12X
  * BRAF V600E
* Patients must be initiating palliative systemic therapy, either on or off a clinical trial

Cohort 4: Paired plasma NGS and ddPCR

* Cohort 4A (CLOSED):

  * Advanced NSCLC, newly diagnosed or with progression following treatment.
  * Biopsy tissue must be available or a biopsy planned and one of the following:

    * Genotyping must have been performed previously
    * Genotyping must be in progress
    * A plan must exist to order genotyping on existing tissue or a planned re-biopsy
  * Patient must not be eligible to enroll in cohort 1A or 2A due to:

    * Not eligible for cohort 1A or 2A
    * Eligible for cohort 1A or 2A but cohort has closed
* Cohort 4B: Undergenotyped NSCLC

  * Advanced NSCLC, newly diagnosed or with progression following treatment.
  * No known targetable genotype on prior tumor genotyping
  * Biopsy planned for tumor genotyping
* Cohort 4C: EGFR-mutant NSCLC with acquired resistance

  * Advanced EGFR-mutant NSCLC with progression on EGFR TKI
  * Biopsy planned for resistance genotyping (e.g. T790M, etc)

Cohort 5: Genotyped KRAS patients starting palliative systemic therapy

* Advanced NSCLC harboring a KRAS exon 2 mutation
* Patients must be initiating new systemic therapy, either on or off a clinical trial

Exclusion Criteria

* Participants who are unable to provide informed consent
* Participants who are 18 years of age or younger
* Participants who are unable to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC and advanced melanoma that are either newly diagnosed, have acquired resistance to kinase inhibitor therapy or have a known targetable mutation and are beginning a new line of therapy.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2014-07-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Plasma Genotyping Assay | 2 years
  We will determine the accuracy of a droplet digital PCR (ddPCR)-based plasma genotyping assay in performing noninvasive tumor genotyping.

SECONDARY OUTCOMES:
Turnaround Time of Plasma Genotyping Assay | 2 years
  The amount of time required to perform this noninvasive genotyping assay.
Early Treatment Failure | 2 years
  The ability of serial quantitative ddPCR-based plasma genotyping to predict early treatment failure in patients initiating a new line of therapy.
Accuracy of Plasma NGS | 2 years
  We will determine the accuracy of plasma NGS in performing noninvasive genotyping compared to tumor NGS and paired ddPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Rotow, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States